CLINICAL TRIAL: NCT05993078
Title: Safety and Efficacy of Immediate Normal Saline Infusion for Stroke After Intravenous Thrombolysis (NS-STAR)
Brief Title: Normal Saline Infusion for Stroke After Intravenous Thrombolysis
Acronym: NS-STAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Affliated Hospital of Jiujiang University (Unknown); Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, Jiayue Ding, Principle investigator, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NS-STAR
Record Dates: First submitted 2023-08-03; First posted 2023-08-15 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Brain Infarct
Keywords: brian infarction; thrombolysis; haemodilution; normal saline
MeSH Terms: conditions — Brain Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NS group (Experimental): The patient will undergo NS 2000ml intravenous infusion immediately after IVT.
  Interventions: Drug: 0.9% NaCl 2000ml
- Control group (Placebo Comparator): The patient will the patients receive an NS 200-400ml after IVT.
  Interventions: Drug: 0.9% NaCl 200-400ml

INTERVENTIONS:
Drug: 0.9% NaCl 2000ml — The patient will undergo NS 2000ml intravenous infusion immediately after IVT. Subsequent therapy is based on Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2018. All of the subjects should be treated in the hospital at least 7 days according to the guidelines for early management of stroke.
  Arms: NS group
Drug: 0.9% NaCl 200-400ml — The patients receive an NS 200-400ml after IVT. Subsequent therapy is based on Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2018. All of the subjects should be treated in the hospital at least 7 days according to the guidelines for early management of stroke.
  Arms: Control group

SUMMARY:
This study aims to explore the safety and efficacy of 0.9% normal saline （NS） infusion on stroke after intravenous thrombolysis (IVT), we decided to conduct this multi-centre randomized controlled trial for the first time. This trial will provide an innovative strategy to facilitate functional independence after stroke administered with IVT. This is a multi-center, randomized controlled two arm (1:1 ratio) clinical trial. The enrolled participators will be divided into the NS group and the control group randomly after confirming as acute ischemic stroke (AIS). In the NS group, the patient will undergo NS 2000ml intravenous infusion immediately after IVT, with the speed of 200ml/h. In the control group, the patient will receive an NS 200-400ml after IVT. The primary efficacy is disability at days 90, as scored by means of the modified Rankin scale (mRS), dichotomized as a favorable outcome (a score of 0-2), or an unfavorable outcome (a score of 3 to 6). The secondary outcomes mainly comprise neurological deficits, disability, imaging and laboratory tests at each follow-up time. The safety outcomes include the cerebral edema at 24-hour post-IVT detected by cranial CT, the 24-hour fluctuation of blood pressure and the cardiac function detected by ultrasonic cardiogram within 3 days after IVT.

ELIGIBILITY:
Inclusion criteria

1. AIS;
2. Age 18-80 years;
3. Prestroke mRS≤1;
4. NIHSS score 0-25;
5. Onset-to-needle time≤4.5 h;
6. Sign the informed consent. Exclusion criteria

(1) Massive infarction, characterized by infarction area larger than 1/3 of the effected middle cerebral artery territory and/or the cerebellum territory presented in admitted computed tomography (CT) or MRI; (2) Intention to undergo endovascular treatment; (3) History of heart failure or pre-IVT BNP≥500pg/ml or having presentations or signs indicating heart failure; (4) Haemorrhage during IVT, including ICH, severe digestive haemorrhage and severe respiratory haemorrhage; (5) Allergy to thrombolysis drugs; (6) Intolerant to thrombolysis due to any reasons and had to terminate thrombolysis; (7) Arterial puncture at a non-compressible site within previous 7 days, major surgery within previous 14 days, sever trauma, gastrointestinal or urinary tract bleeding within previous 21 days; (8) Cerebral infarction or myocardial infarction within previous 3 months, previous intracranial haemorrhage (ICH) including parenchymal haemorrhage, intraventricular haemorrhage, subarachnoid haemorrhage, subdural/external haematoma, etc; (9) Severe brain trauma, intracranial or intraspinal surgery within previous 3 months or known malignant intracranial neoplasm, giant intracranial aneurysm or arteriovenous malformation; (10) Persistent systolic blood pressure≥180mmHg or diastolic blood pressure≥100mmHg; (11) Admitted blood glucose<2.8mmol/L or >22.22mmol/L; (12) Defect in coagulation, for example, current use of oral warfarin with an international normalised ratio>1.7, or prothrombin time>15s, or heparins during the last 48 hours, or use of direct thrombin inhibitors or direct factor Xa inhibitors during the last 48 hours or with an elevated activated partial thromboplastin time; (13) Known defect of platelet or clotting function, platelet count<100×109/L; (14) Stroke mimics, such as seizure and hysteria; (15) Brain haemorrhage identified by CT or MRI; (16) Any terminal illness such that patients would not be expected to survive>1 year; (17) Pregnant women or nursing mother; (18) Poor compliance, or inability to adhere to the trial protocol or follow-up; (19) Participating in other clinical trials within previous 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine of Hebei Province, Cangzhou, Heibei
  - Affiliated Hospital of Jiujiang University, Jiujiang, Jiangxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
We will share study protocol and statistical analysis plan with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: One years after publications.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NS Group | Control Group
Started | 121 | 120
Completed | 121 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NS Group | Control Group | Total
Number analyzed (Participants) | 121 | 120 | 241
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [60.5 to 71] | 66 [60 to 71] | 67 [60 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 86 | 82 | 168
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 121 | 120 | 241

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 90-day Favorable Outcome
Description: Disability on day 90, as scored by means of the modified Rankin scale (mRS), dichotomized as a favorable outcome (a score of 0 to 2), or an unfavorable outcome (a score of 3 to 6). Scores on mRS range from 0 (no symptoms at all) to 6 (death), with higher values reflecting more severe disability or death.
Time Frame: 90 days
Population: One patient in each group was lost to follow-up at 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 120 | 119
Participants | 106 | 93

2. Secondary Outcome: NIHSS Scores at 24 Hours
Description: The National Institutes of Health Stroke Scale (NIHSS), a 15-item scale that measures the level of neurologic impairment. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts (<5, mild impairment; ≥25, very severe neurologic impairment).
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 120
score on a scale | 2 [0 to 4] | 2 [1 to 5]

3. Secondary Outcome: NIHSS Scores on Day 7
Description: as for outcome 2
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 120 | 114
score on scale | 1 [0 to 3] | 1 [0 to 3]

4. Secondary Outcome: mRS on Day 7
Description: Scores on the modified Rankin scale(mRS) range from 0 (no symptoms at all) to 6 (death), with higher values reflecting more severe disability or death.
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 117
score on scale | 1 [0 to 2] | 1 [1 to 3]

5. Secondary Outcome: mRS on Day 30
Description: as for outcome 4
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 120
score on a scale | 1 [0 to 2] | 1 [0 to 2]

6. Secondary Outcome: Number of Participants With Barthel Index 60-100 on Day 30
Description: The Barthel Index represents functional status at follow-up time, the scores of which range from 0 (complete dependence) to 100 (complete independence) measured by several items, including feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfers, and stairs.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 120 | 116
Participants | 108 | 104

7. Secondary Outcome: Number of Participants With Barthel Index 60-100 on Day 90
Description: as for outcome 6
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 118 | 114
Participants | 111 | 105

8. Secondary Outcome: Number of Pariticipants With Early Neurological Deterioration (END, △NIHSS≥2)
Description: Early neurological deterioration (END) indicates an increase of ≥2 in the NIHSS score within 24 hours after IVT, and the deterioration is not caused by intracranial hemorrhage that is confirmed by cranial CT. The National Institutes of Health Stroke Scale (NIHSS), a 15-item scale that measures the level of neurologic impairment. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 120 | 120
Participants | 10 | 25

9. Secondary Outcome: Number of Participants With Early Neurological Deterioration (END, △NIHSS≥4)
Description: Early neurological deterioration (END) indicates an increase of ≥4 in the NIHSS score within 24 hours after IVT, and the deterioration is not caused by intracranial hemorrhage that is confirmed by cranial CT. The National Institutes of Health Stroke Scale (NIHSS), a 15-item scale that measures the level of neurologic impairment. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 120 | 120
Participants | 8 | 19

10. Secondary Outcome: Imaging Infarction Volume at 24 Hours
Description: Cranial computed tomography (CT) scans are performed before IVT and 24 hours after randomization. The infarction area is confirmed using CT maps and the infarction volume is calculated by 3D-Slicer (Version4.6.2, https://www.slicer.org/).
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 118
ml | 0.21 [0 to 2.52] | 0.31 [0 to 1.82]

11. Secondary Outcome: Blood Pressure at 24 Hours
Description: Blood pressure, including systolic blood pressure (SBP) and diastolic blood pressure (DBP), is monitored at 24 hours after randomization.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 120
mmHg
  systolic pressure | 142 [133 to 158] | 135 [123 to 148]
  diastolic pressure | 79 [72 to 87] | 77 [71 to 83]

12. Secondary Outcome: Ejection Fraction
Description: Ejection fraction was assessed by ultrasonic cardiogram within 72 hours after randomization.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 111 | 92
percentage | 63 [62 to 64] | 63 [60 to 64]

13. Secondary Outcome: Death Rate
Description: Death rate within 90 days after randomization.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 120 | 119
Participants | 2 | 5

14. Secondary Outcome: Number of Paricipants With Intracaranial Hemorrhage
Description: Intracaranial hemorrhage confirmed by cranial CT within 7 days after randomization.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 120
Participants | 7 | 3

15. Secondary Outcome: Number of Participants With Symptomatic Intracranial Hemorrhage
Description: Symptomatic intracranial hemorrhage indicates NIHSS deterioration≥2 scores in combination with intracranial hemorrhage on CT scan without other causes for the deterioration within 7 days after randomization.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 121 | 120
Participants | 2 | 0

16. Secondary Outcome: Neutrophil-to-lymphocyte Ratio (NLR)
Description: Peripheral blood inflammatory indices, neutrophil-to-lymphocyte ratio (NLR),24-48 hours after randomization.
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 114 | 110
ratio | 2.75 [1.96 to 3.87] | 2.63 [1.94 to 3.81]

17. Secondary Outcome: Platelet-to-lymphocyte (PLR)
Description: Peripheral blood inflammatory indices, platelet-to-lymphocyte (PLR) at 24-48 hours after randomization.
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 114 | 110
ratio | 135.70 [99.78 to 158.35] | 128.11 [100.71 to 159.30]

18. Secondary Outcome: SII
Description: Peripheral blood inflammatory indices, (platelet✖neurophil)/lymphocyte (SII) at 24-48 hours after randomization.
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 114 | 110
ratio | 527.05 [382.92 to 833.79] | 531.51 [426.70 to 796.46]

19. Secondary Outcome: S100-β
Description: Laboratory examinations, peripehral S100-β at 24-48 hours after randomization.
Time Frame: 24-48 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 110 | 88
ng/ml | 2.17 (5.82) | 1.22 (2.19)

20. Secondary Outcome: Myeloperoxidase (MPO)
Description: Laboratory examinations, peripheral myeloperoxidase (MPO) at 24-48 hours after randomization.
Time Frame: 24-48 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 110 | 88
pg/ml | 52746.41 (35023.82) | 53902.99 (47152.39)

21. Secondary Outcome: Brain Derived Neurotrophic Factor (BDNF)
Description: Laboratory examinations, brain derived neurotrophic factor (BDNF)at 24-48 hours after randomization.
Time Frame: 24-48 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | NS Group | Control Group
Number analyzed (Participants) | 107 | 77
pg/ml | 1019.59 (810.89) | 999.6 (817.42)

ADVERSE EVENTS:
Time Frame: through 90 days
Description: Adverse events include all death, serious adverse events and other adverse events. Serous adverse events comprise (1) fatal; (2) life-threatening; (3) causing or prolonging hospitalization; (4) disability or organ function impairment. Other adverse events include acute heart failure, hypertensive crisis, edema (such as severe cerebral edema, pulmonary edema, limb edema and water intoxication) and other severe complications.
Arm/Group | NS Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/121 | 5/120
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/120
Other Adverse Events (participants affected / at risk) | 0/121 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT05993078/Prot_SAP_000.pdf